CLINICAL TRIAL: NCT06695273
Title: Using Retinal Photograph Based AI to Predict Incident Coronary Heart Disease
Acronym: DeepCHD Plus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Tien Yin Wong, Professor, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: DeepCHD Plus
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Coronary Heart Disease (CHD)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-Assisted Group (AI Group) (Experimental): Physicians receive CHD probability estimates from an AI model based on retinal photographs. The AI tool provides individualized CHD probabilities, leveraging retinal biomarkers associated with cardiovascular risk.
  Interventions: Diagnostic Test: AI-derived probability of coronary heart disease.
- Guideline-Based Group (Guideline Group) (Active Comparator): Physicians use a PCE calculator to calculate the 10 year ASCVD risk. This approach aligns with current clinical guidelines to assist in decision-making.
  Interventions: Diagnostic Test: PCEs derived ASCVD risk

INTERVENTIONS:
Diagnostic Test: AI-derived probability of coronary heart disease. — Physician readers will be assisted with AI-derived probability of coronary heart disease. The AI tool provides individualized obstructive CHD probabilities and diagnosis, leveraging retinal biomarkers associated with cardiovascular risk.
  Arms: AI-Assisted Group (AI Group)
Diagnostic Test: PCEs derived ASCVD risk — Physicians use a PCEs to calculate the probability of 10 year ASCVD risk. This approach aligns with current clinical guidelines to assist in decision-making.
  Arms: Guideline-Based Group (Guideline Group)

SUMMARY:
To determine whether an integrated retinal AI decision support can improve predictive accuracy of coronary heart disease (CHD), the investigators are conducting a randomized controlled study of AI guided prediction of CHD compared to clinical prediction by physicians (e.g., usingPCEs), both using clinical intuition as baseline.

DETAILED DESCRIPTION:
This is a randomized controlled trial (RCT) evaluating the effectiveness of an AI-based decision support tool in CHD risk prediction and decision making by physicians. Prospective cohort study participant cases will be randomly assigned to either guideline group (e.g., PCEs) or AI group after baseline assessment (clinical intuition):

There are three settings: (1) Clinical Intuition (baseline assessment) Physicians' make decision about prevention strategy initiation (e.g., statin initiation) without any external assistance. Assessment relies solely on the physician's clinical judgment and experience. (2) Guideline-Based Group (Guideline Group) Physicians use a PCE table to calculate the 10 year ASCVD risk. This approach aligns with current clinical guidelines to assist in decision-making. (3) AI-Assisted Group (AI Group) Physicians receive CHD probability estimates from an AI model based on retinal photographs. The AI tool provides individualized obstructive CHD probabilities, leveraging retinal biomarkers associated with cardiovascular risk.

Primary Objective To evaluate whether AI-guided decision support could improves diagnostic accuracy of CHD to a greater extent than standard clinical assessments, both compared to clinical intuition. The accuracy could be assessed by the extent of prevention initiation (e.g., prescribing statins) corresponding with actual CHD outcomes observed.

Secondary Objective To assess whether AI-guided decision support reduces the time required to complete CHD assessments and decision making.

Participants, Readers and Randomization:

Participants: Participants in prospective cohort studies, with 10-year follow up.

Readers: Physicians performing evaluations of CHD probability and make primary prevention recommendations.

Randomization: Participants will be randomized into one of the groups (PCEs or AI) after clinical assessment at baseline using block randomization to ensure balanced group sizes.

ELIGIBILITY:
Inclusion criteria:

* Individuals without uncontrolled vascular risk factors
* Age range: 40-75 years old
* Can accept and cooperate with the examination and potential follow-up work after being selected for clinical trials

Exclusion criteria:

* Severe lung disease and cancer or surgery patients
* Statin user or pre-existing cardiovascular disease
* Individuals with severe liver and kidney dysfunction and electrolyte imbalance

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1570 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy | Through study completion, an average of 1 week
  To evaluate whether AI-guided decision support could improves diagnostic accuracy of CHD to a greater extent than standard clinical assessments, both compared to clinical intuition. The accuracy could be assessed by the degree to which prevention initiation (e.g., prescribing statins) align with actual CHD outcomes observed.

CONTACTS AND LOCATIONS:
Overall Officials: Tien Yin Wong, Principal Investigator — Tsinghua University